CLINICAL TRIAL: NCT05661656
Title: Role of Catheter Guided Intra-arterial Chemo-infusion in Breast Cancer.
Brief Title: Catheter Guided Chemo-infusion in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed ahmed abdel wahab, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: catheter guided chemo-infusion
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Adult female had stage III,IV breast cancer with no prior chemotherapy, radiotherapy, or definitive surgical therapy for breast cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced breast cancer patients (Experimental): Tumors are staged according to the criteria of the Union for International Cancer Control (UICC). Tumor volume was determined by mammography or magnetic resonance imaging (MRI). Patients will be cannulated via the femoral artery. Then, a 4F fixed-curve catheter (Cobra catheter, Cook Corporation, Bloomington) was advanced to the ipsilateral subclavian artery. Digital subtraction angiography (DSA) was performed to determine tumor arterial blood supply. Super selection of the internal mammary artery done by micro-catheter. Chemo-infusion was decided by the major feeding artery. The intra-arterial chemoinfusion regimen consisted of docetaxel 75 mg/m2 and epirubicin 50 mg/m2 in 200 mL of normal saline and 5% glucose; the drugs were slowly infused via the catheter over at least 15 minutes. Intraarterial infusion was performed once every 3 weeks on average.
  Interventions: Procedure: Intra-arterial chemoinfusion of breast cancer

INTERVENTIONS:
Procedure: Intra-arterial chemoinfusion of breast cancer — Patients will be cannulated via the femoral artery. Then, a 4F fixed-curve catheter (Cobra catheter, Cook Corporation, Bloomington) was advanced to the ipsilateral subclavian artery. Digital subtraction angiography (DSA) was performed to determine tumor arterial blood supply. Super selection of the internal mammary artery done by micro-catheter. Chemo-infusion was decided by the major feeding artery. The intra-arterial chemoinfusion regimen consisted of docetaxel 75 mg/m2 and epirubicin 50 mg/m2 in 200 mL of normal saline and 5% glucose; the drugs were slowly infused via the catheter over at least 15 minutes. Intraarterial infusion was performed once every 3 weeks on average.

SUMMARY:
In the present prospective study, we will analyze the outcome of image-guided delivery of intra-arterially infused chemotherapeutic drugs for patients with breast cancer in III, IV stages.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies affecting women worldwide, and its incidence has seen a steady increase over the years with the involvement of women at a much younger age, which poses a serious health threat to women and has a staggering global impact.

Lymph node and hematogenous metastasis occurs at the early stage of breast cancer and is the principal cause of mortality of breast cancer patients.

Surgical resection is the most effective method for the treatment of breast cancer, and neoadjuvant chemotherapy reduces the risk of disease recurrence and death in women who have operable breast cancer.

For patients with inoperable breast cancer, neoadjuvant chemotherapy reduces tumor bulk and tumor stage, thereby increasing the chance of surgical resection and reducing postoperative tumor recurrence and metastasis.

Local or regional chemotherapy is an alternative for reducing metastatic lesions and increasing patient survival .Intra-arterial infusion chemotherapy (chemoinfusion), a form of regional chemotherapy, has been used in the treatment of gastrointestinal tumors, liver cancer, and pancreatic cancer.

In the present prospective study, we will analyze the outcome of image-guided delivery of intra-arterially infused chemotherapeutic drugs for patients with breast cancer in III, IV stages.

ELIGIBILITY:
Inclusion Criteria:

* Adult female had stage III,IV breast cancer.
* Female had received no prior chemotherapy, radiotherapy, or definitive surgical therapy for breast cancer.
* Patient had adequate organ function.

Exclusion Criteria:

* Patients known to have absolute contraindications for contrast.
* Patient known to have systemic organ failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Lesion size after chemotherapy | 3 weeks
  Patient will be evaluated 3 weeks after the second intra-arterial chemo infusion. If the primary lesion and the involved lymph nodes shrunken markedly in volume and skin and muscle involvement improved noticeably, patients were assigned to undergo surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Abdelwahab, MSc, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Veronesi U, Boyle P, Goldhirsch A, Orecchia R, Viale G. Breast cancer. Lancet. 2005 May 14-20;365(9472):1727-41. doi: 10.1016/S0140-6736(05)66546-4. PMID 15894099
- [Result] Vinh-Hung V, Verschraegen C, Promish DI, Cserni G, Van de Steene J, Tai P, Vlastos G, Voordeckers M, Storme G, Royce M. Ratios of involved nodes in early breast cancer. Breast Cancer Res. 2004;6(6):R680-8. doi: 10.1186/bcr934. Epub 2004 Oct 6. PMID 15535850
- [Result] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097